CLINICAL TRIAL: NCT00364975
Title: Development of Gourmet Healthy Cooking Workshop for Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was not funded
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 31150906-HMO-CTIL
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2006-08

CONDITIONS: Breast Cancer
Keywords: gourmet healthy cooking; quality of life; adjuvant chemotherapy; weight; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Body Weight

INTERVENTIONS:
Behavioral: gourmet cooking workshop

SUMMARY:
Subjects that participate in the practical workshop will improve their metabolic indexes, control their weight and improve their quality of life, in contrast to the participants that will take part in the nutritional consulting sessions

DETAILED DESCRIPTION:
Participants will be randomly assigned to a dietary consultation-only control group or to a gourmet medical cooking workshop. The workshop will consist of 6 lessons with the following lessons: introduction, caloric density of food, fats, vegetable and fruits, Whole grains and legumes, Healthy desserts . All the lessons will start with half an hour theoretical introduction, followed by a 2.5 hours "hands on" session under supervision of a medical chef. The study population will include women receiving adjuvant chemotherapy for breast cancer. 72 patients will be recruited and will be randomly divided into two groups: an intervention group of 36 will commence the workshop during 2007 and a control group of 36 who will take part in dietitian consulting sessions only.

ELIGIBILITY:
Inclusion Criteria:

* Adjuvant chemotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Primary: We expect to see change in the following outcomes: the patient's metabolic state, the patient's weight, body composite, patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: berry elliot, md, Principal Investigator — hadassah univercity hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel